CLINICAL TRIAL: NCT00304031
Title: Phase III Trial Comparing Conventional Adjuvant Temozolomide With Dose-Intensive Temozolomide in Patients With Newly Diagnosed Glioblastoma
Brief Title: Radiation Therapy (RT) and Temozolomide (TMZ) in Treating Patients With Newly Diagnosed Glioblastoma or Gliosarcoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); European Organisation for Research and Treatment of Cancer - EORTC (Network); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0525; CDR0000465183; EORTC-26052; EORTC-22053; NCI-2009-00731 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Results first posted 2014-04-30 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2020-05

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Conventional adjuvant TMZ (Active Comparator): Concurrent radiation therapy with concurrent temozolomide (75 mg/m2) up to 49 doses. Starting four weeks after completion of RT, 100mg/m2 adjuvant temozolomide days 1 to 5 of 28 day cycle.
  Interventions: Drug: Concurrent temozolomide; Radiation: Concurrent radiation therapy; Drug: 100mg/m2 adjuvant temozolomide days 1 to 5 of 28 day cycle
- Dose-dense adjuvant TMZ (Experimental): Concurrent radiation therapy (RT) with concurrent temozolomide (75 mg/m2) up to 49 doses. Starting four weeks after completion of RT, 75mg/m2 adjuvant temozolomide days 1-21 of 28 day cycle.
  Interventions: Drug: Concurrent temozolomide; Radiation: Concurrent radiation therapy; Drug: 75mg/m2 adjuvant temozolomide days 1-21 of 28 day cycle
- No adjuvant TMZ (not randomized ) (Other): Concurrent radiation therapy (RT) with concurrent temozolomide (75 mg/m2) up to 49 doses. Not randomized to either adjuvant TMZ arm.
  Interventions: Drug: Concurrent temozolomide; Radiation: Concurrent radiation therapy

INTERVENTIONS:
Drug: Concurrent temozolomide — Daily oral temozolomide (75 mg/m2) up to 49 doses.
Radiation: Concurrent radiation therapy — 60 Gy in 2 Gy fractions
Drug: 100mg/m2 adjuvant temozolomide days 1 to 5 of 28 day cycle — Oral temozolomide on days 1-5 of a 28-day cycle. Dose starts at 150mg/m2 for first cycle, increases to 200mg/m2 for subsequent cycles if no unacceptable toxicity. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients with responding disease may receive up to 6 more courses of temozolomide.
  Arms: Conventional adjuvant TMZ
Drug: 75mg/m2 adjuvant temozolomide days 1-21 of 28 day cycle — Oral temozolomide on days 1-21 of a 28-day cycle. Dose starts at 75mg/m2 for first cycle, increases to 100mg/m2 for subsequent cycles if no unacceptable toxicity. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients with responding disease may receive up to 6 more courses of temozolomide.
  Arms: Dose-dense adjuvant TMZ

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving radiation therapy together with temozolomide may kill more tumor cells. It is not yet known which schedule of temozolomide when given together with radiation therapy is more effective in treating glioblastoma or gliosarcoma.

PURPOSE: This randomized phase III trial is studying two different schedules of temozolomide to compare how well they work when given together with radiation therapy in treating patients with newly diagnosed glioblastoma or gliosarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine if dose-intensifying (increasing the "dose-density") the adjuvant temozolomide component of the chemoradiation treatment enhances treatment efficacy as measured by overall survival of patients with newly diagnosed glioblastoma or gliosarcoma.

Secondary

* Determine if dose-intensifying the adjuvant temozolomide component of the chemoradiation treatment enhances treatment efficacy as measured by progression-free survival.
* Determine in patients with unmethylated MGMT (O-6-methylguanine-DNA methyltransferase) if dose-intensifying the adjuvant temozolomide component of the chemoradiation treatment enhances treatment efficacy (overall and progression-free survival) compared with patients receiving conventional temozolomide dosing.
* Determine in patients with methylated MGMT if dose-intensifying the adjuvant temozolomide component of the chemoradiation treatment enhances treatment efficacy (overall and progression-free survival) compared with patients receiving conventional temozolomide dosing.
* Determine if there is an association between tumor MGMT gene methylation status and treatment response.
* Compare and record the toxicities of the conventional and dose-intense chemotherapy regimens.
* Evaluate whether 6-month progression-free survival is associated with overall survival.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to recursive partitioning analysis class (III vs IV vs V), MGMT gene methylation status (methylated vs nonmethylated vs indeterminate), and radiotherapy criteria used (standard vs revised European).

After completion of study treatment, patients are followed every 3 months for 1 year, every 4 months for 2 years, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion criteria:

1. Histopathologically proven diagnosis of glioblastoma. Since gliosarcoma is a variant of glioblastoma, gliosarcoma is also an eligible diagnosis.
2. Patients must have at least 1 block of tissue available for analysis of MGMT status; fresh frozen tumor tissue acquisition is encouraged.
3. Diagnosis must be established by open biopsy or tumor resection. Patients who have only had a stereotactic biopsy are not eligible.
4. The tumor must have a supratentorial component.
5. Patients must have recovered from the effects of surgery, postoperative infection, and other complications before study registration.
6. A diagnostic contrast-enhanced magnetic resonance imaging (MRI) or computerized tomography (CT) scan (if MRI is not available) of the brain must be performed preoperatively and postoperatively. The postoperative scan must be done within 28 days of registration and prior to the initiation of radiotherapy. Preoperative and postoperative scans must be the same type. If CT scans were performed perioperatively, a CT and an MRI should be performed before randomization.

   6.1. Patients unable to undergo MRI imaging because of non-compatible devices can be enrolled, provided pre- and post-operative contrast-enhanced CT scans are obtained and are of sufficient quality.
7. Therapy must begin ≤ 5 weeks after the most recent brain tumor surgery.
8. History/physical examination within 14 days prior to study registration.
9. Neurologic examination within 14 days prior to study registration.
10. Documentation of steroid doses within 14 days prior to study registration and stable or decreasing steroid dose within 5 days prior to registration.
11. Karnofsky performance status of ≥ 60.
12. Age ≥ 18 years.
13. Complete blood count (CBC)/differential obtained within 14 days prior to study registration, with adequate bone marrow function as defined below: 13.1 Absolute neutrophil count (ANC) ≥ 1500 cells/mm3. 13.2 Platelets ≥ 100,000 cells/mm3. 13.3 Hemoglobin ≥ 10 g/dl. (Note: The use of transfusion or other intervention to achieve Hgb ≥ 10 g/dl is acceptable.)
14. Adequate renal function, as defined below:

    14.1 Blood urea nitrogen (BUN) ≤ 25 mg/dl within 14 days prior to study registration 14.2 Creatinine ≤ 1.7 mg/dl within 14 days prior to study registration
15. Adequate hepatic function, as defined below:

    15.1 Bilirubin ≤ 2.0 mg/dl within 14 days prior to study registration 15.2 Alanine aminotransferase (ALT) ≤ 3 x normal range within 14 days prior to study registration 15.3 Aspartate aminotransferase (AST) ≤ 3 x normal range within 14 days prior to study registration
16. Patients must sign a study-specific informed consent prior to study registration.

    If the patient's mental status precludes his/her giving informed consent, written informed consent may be given by the responsible family member.
17. For females of child-bearing potential, negative serum pregnancy test within 72 hours prior to starting temozolomide.
18. Women of childbearing potential and male participants must practice adequate

Exclusion criteria:

1. Prior invasive malignancy (except for non-melanomatous skin cancer) unless disease free for ≥ 3 years. (For example, carcinoma in situ of the breast, oral cavity, and cervix are all permissible).
2. Recurrent or multifocal malignant gliomas
3. Metastases detected below the tentorium or beyond the cranial vault.
4. Prior chemotherapy or radiosensitizers for cancers of the head and neck region; note that prior chemotherapy for a different cancer is allowable. Prior use of Gliadel wafers or any other intratumoral or intracavitary treatment are not permitted. See Section 1.
5. Prior radiotherapy to the head or neck (except for T1 glottic cancer), resulting in overlap of radiation fields.
6. Severe, active co-morbidity, defined as follows:

   * 6.1. Unstable angina and/or congestive heart failure requiring hospitalization.
   * 6.2. Transmural myocardial infarction within the last 6 months.
   * 6.3. Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration.
   * 6.4. Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration.
   * 6.5. Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol.
   * 6.6. Acquired Immune Deficiency Syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive.
   * 6.7. Major medical illnesses or psychiatric impairments that in the investigator's opinion will prevent administration or completion of protocol therapy.
   * 6.8. Active connective tissue disorders, such as lupus or scleroderma, that in the opinion of the treating physician may put the patient at high risk for radiation toxicity.
7. Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.
8. Pregnant or lactating women, due to possible adverse effects on the developing fetus or infant due to study drug;
9. Prior allergic reaction to temozolomide.
10. Patients treated on any other therapeutic clinical protocols within 30 days prior to study entry or during participation in the study.
11. No tissue provided for histopathologic central review and MGMT status.
12. Tissue provided by stereotactic biopsy method.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1173 (Actual)
Dates: Start 2006-01; Primary Completion 2011-02 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark R. Gilbert, MD, Principal Investigator — M.D. Anderson Cancer Center; Minesh P. Mehta, MD, Study Chair — University of Wisconsin, Madison; Roger Stupp, MD, Study Chair — Centre Hospitalier Universitaire Vaudois
Locations (351):
- United States (341):
  - Fairbanks Cancer Treatment Center at Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Arizona Oncology Services Foundation, Phoenix, Arizona
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Arizona Oncology - Tucson, Tucson, Arizona
  - Auburn Radiation Oncology, Auburn, California
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Radiation Oncology Centers - Cameron Park, Cameron Park, California
  - Mercy Cancer Center at Mercy San Juan Medical Center, Carmichael, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente Medical Center - Los Angeles, Los Angeles, California
  - Radiation Oncology Center - Roseville, Roseville, California
  - Radiological Associates of Sacramento Medical Group, Incorporated, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Solano Radiation Oncology Center, Vacaville, California
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - Poudre Valley Radiation Oncology, Fort Collins, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Eugene M. and Christine E. Lynn Cancer Institute at Boca Raton Community Hospital - Main Campus, Boca Raton, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Integrated Community Oncology Network at Southside Cancer Center, Jacksonville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Baptist Medical Center South, Jacksonville, Florida
  - Integrated Community Oncology Network, Jacksonville Beach, Florida
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - Integrated Community Oncology Network - Orange Park, Orange Park, Florida
  - Florida Cancer Center - Palatka, Palatka, Florida
  - Flagler Cancer Center, Saint Augustine, Florida
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - John B. Amos Cancer Center, Columbus, Georgia
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - InterCommunity Cancer Center of Western Illinois, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Valley Cancer Center, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Radiation Oncology Associates Southwest, Fort Wayne, Indiana
  - Parkview Regional Cancer Center at Parkview Health, Fort Wayne, Indiana
  - Central Indiana Cancer Centers - East, Indianapolis, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Kansas City Cancer Centers - Southwest, Overland Park, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - DeCesaris Cancer Institute at Anne Arundel Medical Center, Annapolis, Maryland
  - St. Agnes Hospital Cancer Center, Baltimore, Maryland
  - Union Hospital Cancer Program at Union Hospital, Elkton, Maryland
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Alexandria, Minnesota
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Independence Regional Health Center, Independence, Missouri
  - St. John's Regional Medical Center, Joplin, Missouri
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - St. Joseph Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Parvin Radiation Oncology, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Kansas City Cancer Centers - South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Dartmouth - Hitchcock Concord, Concord, New Hampshire
  - Kingsbury Center for Cancer Care at Cheshire Medical Center, Keene, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - St. Barnabas Medical Center Cancer Center, Livingston, New Jersey
  - Frederick R. and Betty M. Smith Cancer Treatment Center, Sparta, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - New York Methodist Hospital, Brooklyn, New York
  - Monter Cancer Center of the North Shore-LIJ Health System, Lake Success, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Hudson Valley Oncology Associates, Poughkeepsie, New York
  - Lipson Cancer and Blood Center at Rochester General Hospital, Rochester, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Wilmed Radiation Oncology Services, Wilson, North Carolina
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Cleveland Clinic Cancer Center at Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Cleveland Clinic Cancer Center, Independence, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Cancer Research UK Medical Oncology Unit at Churchill Hospital & Weatherall Institute of Molecular Medicine - Oxford, Salem, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Willamette Valley Cancer Center - Eugene, Eugene, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center and Children's Hospital, Portland, Oregon
  - Salem Hospital Regional Cancer Care Services, Salem, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - Dale and Frances Hughes Cancer Center at Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Riddle Memorial Hospital Cancer Center, Media, Pennsylvania
  - Upper Delaware Valley Cancer Center, Milford, Pennsylvania
  - Intercommunity Cancer Center, Monroeville, Pennsylvania
  - Alle-Kiski Medical Center, Natrona Heights, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Frankford Hospital Cancer Center - Torresdale Campus, Philadelphia, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - Somerset Oncology Center, Somerset, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - CCOP - Main Line Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Thompson Cancer Survival Center West, Knoxville, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Thompson Cancer Survival Center at Methodist, Oak Ridge, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - Texas Oncology, PA at Texas Cancer Center Dallas Southwest, Dallas, Texas
  - Klabzuba Cancer Center at Harris Methodist Fort Worth Hospital, Fort Worth, Texas
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Texas Oncology, PA at Texas Cancer Center - Sherman, Sherman, Texas
  - Texas Oncology, PA at Texas Oncology Cancer Center Sugar Land, Sugar Land, Texas
  - American Fork Hospital, American Fork, Utah
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Norris Cotton Cancer Center - North, Saint Johnsbury, Vermont
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Sentara Cancer Institute at Sentara Norfolk General Hospital, Norfolk, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - St. Joseph Cancer Center, Bellingham, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Cascade Cancer Center at Evergreen Hospital Medical Center, Kirkland, Washington
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Theda Care Cancer Institute, Appleton, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Community Memorial Hospital Cancer Care Center, Menomonee Falls, Wisconsin
  - Regional Cancer Center at Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Door County Cancer Center at Door County Memorial Hospital, Sturgeon Bay, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
- Canada (10):
  - Tom Baker Cancer Centre - Calgary, Calgary, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Ottawa Hospital Regional Cancer Centre - General Campus, Ottawa, Ontario
  - Cancer Care Program at Thunder Bay Regional Health Sciences, Thunder Bay, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - McGill Cancer Centre at McGill University, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan

REFERENCES:
- [Result] Aldape KD, Wang M, Sulman EP, et al.: RTOG 0525: molecular correlates from a randomized phase III trial of newly diagnosed glioblastoma. [Abstract] J Clin Oncol 29 (Suppl 15): A-LBA2000, 2011.
- [Result] Armstrong TS, Wefel JS, Wang M, et al.: Clinical utility of neurocognitive function (NCF), quality of life (QOL), and symptom assessment as prognostic factors for survival and measures of treatment effects on RTOG 0525. [Abstract] J Clin Oncol 29 (Suppl 15): A-2016, 2011.
- [Result] Wang M, Dignam JJ, Won M, Curran W, Mehta M, Gilbert MR. Variation over time and interdependence between disease progression and death among patients with glioblastoma on RTOG 0525. Neuro Oncol. 2015 Jul;17(7):999-1006. doi: 10.1093/neuonc/nov009. Epub 2015 Feb 16. PMID 25688120
- [Result] Aldape KD, Jones G, Wang M, et al.: MGMT methylation testing in RTOG 0525: A phase III trial of newly diagnosed glioblastoma. [Abstract] J Clin Oncol 27 (Suppl 15): A-2051, 2009.
- [Result] Gilbert MR, Wang M, Aldape KD, Stupp R, Hegi ME, Jaeckle KA, Armstrong TS, Wefel JS, Won M, Blumenthal DT, Mahajan A, Schultz CJ, Erridge S, Baumert B, Hopkins KI, Tzuk-Shina T, Brown PD, Chakravarti A, Curran WJ Jr, Mehta MP. Dose-dense temozolomide for newly diagnosed glioblastoma: a randomized phase III clinical trial. J Clin Oncol. 2013 Nov 10;31(32):4085-91. doi: 10.1200/JCO.2013.49.6968. Epub 2013 Oct 7. PMID 24101040
- [Derived] Bell EH, Pugh SL, McElroy JP, Gilbert MR, Mehta M, Klimowicz AC, Magliocco A, Bredel M, Robe P, Grosu AL, Stupp R, Curran W Jr, Becker AP, Salavaggione AL, Barnholtz-Sloan JS, Aldape K, Blumenthal DT, Brown PD, Glass J, Souhami L, Lee RJ, Brachman D, Flickinger J, Won M, Chakravarti A. Molecular-Based Recursive Partitioning Analysis Model for Glioblastoma in the Temozolomide Era: A Correlative Analysis Based on NRG Oncology RTOG 0525. JAMA Oncol. 2017 Jun 1;3(6):784-792. doi: 10.1001/jamaoncol.2016.6020. PMID 28097324

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Sites were required to submit participant tumor tissue for central histologic review and MGMT (O-6-methylguanine-DNA methyltransferase) status determination in order for registered participants to continue on the study. Of 1173 participants initially registered, 1125 participants met these requirements and started protocol treatment.
Groups:
- No Adjuvant TMZ (Not Randomized): Concurrent radiation therapy (RT) with concurrent temozolomide (TMZ) (75 mg/m2) up to 49 doses. Not randomized to either adjuvant TMZ arm.
Period: Concomitant RT+TMZ (Pre-randomization)
Arm/Group | No Adjuvant TMZ (Not Randomized) | Conventional Adjuvant TMZ | Dose-dense Adjuvant TMZ
Started | 1125 (All participants registered to concomitant treatment; randomized after completing this treatment.) | 0 (Participants were not randomized to adjuvant TMZ until after completion of concomitant treatment.) | 0 (Participants were not randomized to adjuvant TMZ until after completion of concomitant treatment.)
Eligible Pre-randomization Population | 1125 | 0 | 0
Eligible Pre-randomization Follow-up (Eligible pre-randomization participants with any follow-up data.) | 1120 | 0 | 0
Completed | 833 (These participants completed concomitant treatment and met requirements for randomization.) | 0 | 0
Not Completed | 292 | 0 | 0
Not completed — Ineligible due to insufficient tissue | 144 | 0 | 0
Not completed — Disease progression | 48 | 0 | 0
Not completed — Patient refusal | 19 | 0 | 0
Not completed — Death | 18 | 0 | 0
Not completed — Physician preference | 15 | 0 | 0
Not completed — Toxicity | 10 | 0 | 0
Not completed — Other complicating disease | 1 | 0 | 0
Not completed — Other, not otherwise specified | 37 | 0 | 0
Period: Randomization to Adjuvant TMZ Arm
Arm/Group | No Adjuvant TMZ (Not Randomized) | Conventional Adjuvant TMZ | Dose-dense Adjuvant TMZ
Started (Participants who met requirements after concomitant treatment were randomized to an adjuvant arm.) | 0 | 411 | 422
Eligible Population | 0 | 411 | 420
Unmethylated MGMT Population (Eligible participants determined to have unmethylated MGMT.) | 0 | 254 | 262
Methylated MGMT Population (Eligible participants determined to have methylated MGMT.) | 0 | 122 | 122
Quality of Life Population (Eligible participants who consented to the quality of life study component, offered after 07-12-2007) | 0 | 96 | 95
Completed | 0 | 411 (Randomized participants contributing data to results are considered to have completed the study.) | 420 (Randomized participants contributing data to results are considered to have completed the study.)
Not Completed | 0 | 0 | 2
Not completed — No follow-up collected | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Eligible patients who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | No Adjuvant TMZ (Not Randomized ) | Conventional Adjuvant TMZ | Dose-dense Adjuvant TMZ | Total
Number analyzed (Participants) | 292 | 411 | 422 | 1125
Age, Continuous [Median (Full Range); unit: years] | 60.5 [22 to 87] | 57 [22 to 84] | 58 [21 to 84] | 58 [21 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 172 | 185 | 483
  Male | 166 | 239 | 237 | 642

OUTCOME MEASURES:

1. Primary Outcome: Median Overall Survival Time
Description: Overall survival time is defined as time from registration/randomization to the date of death from any cause. Overall survival rates are estimated by the Kaplan-Meier method. Patients last known to be alive are censored at the date of last contact. Analysis occurred after 647 deaths were reported.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 4.4 years.
Population: Randomized eligible patients.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Conventional Adjuvant TMZ: Concurrent radiation therapy with concurrent temozolomide (TMZ) (75 mg/m2) up to 49 doses. Starting four weeks after completion of RT, 100mg/m2 adjuvant temozolomide days 1 to 5 of 28 day cycle.
Arm/Group | Conventional Adjuvant TMZ | Dose-dense Adjuvant TMZ
Number analyzed (Participants) | 411 | 420
months | 16.6 [14.9 to 18.0] | 14.9 [13.7 to 16.5]
Statistical Analysis 1: Comparison: Conventional Adjuvant TMZ vs Dose-dense Adjuvant TMZ; This study was looking for a 20% reduction in hazard rate: null hypothesis (conventional arm): Median survival time (MST) = 14.0 mo.; alternative hypothesis (dose-dense arm): MST= 17.5 mo. A one-sided log-rank test at a significance level of 0.025 would have 80% power to detect this difference with a sample size of 750 patients (647 deaths were required for the final analysis); Test type: Superiority or Other; p = 0.63, Log Rank — One-sided; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.88 to 1.20] — Reference level = Conventional adjuvant TMZ

2. Secondary Outcome: Median Progression-free Survival (PFS) Time
Description: Progression is defined as greater than 25% increase in tumor area (two diameters) provided that the patient has not had his/her dose of steroids decreased since the last evaluation period. Progression-free survival time is defined as time from registration to the date of first progression, death, or last known follow-up (censored). Progression-free survival rates are estimated using the Kaplan-Meier method. A concomitant decrease in steroid dose will rule out a progression designation during the first 2 months after completion of radiation therapy. Analysis occurred after 647 deaths were reported.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 4.4 years.
Population: Randomized eligible patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Conventional Adjuvant TMZ | Dose-dense Adjuvant TMZ
Number analyzed (Participants) | 411 | 420
months | 5.5 [4.7 to 6.1] | 6.7 [6.2 to 7.7]
Statistical Analysis 1: Comparison: Conventional Adjuvant TMZ vs Dose-dense Adjuvant TMZ; Test type: Superiority; p = 0.06, Log Rank — Two-side significance level = 0.05; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.75 to 1.00] — Reference level = Conventional adjuvant TMZ

3. Secondary Outcome: Median Overall Survival Time by MGMT Status
Description: Overall survival time is defined as time from randomization to the date of death from any cause. Overall survival rates are estimated by the Kaplan-Meier method. Patients last known to be alive are censored at the date of last contact. Tumor tissue submitted at baseline was analyzed to determine MGMT (O[6]-methylguanine-DNA methyltransferase) promoter methylation status (methylated / unmethylated). Analysis occurred after 647 deaths were reported.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 4.4 years.
Population: MGMT status was not available for all randomized eligible participants. Therefore, data was only available from 376/411 on the conventional arm and 384/420 on the dose-dense arm.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Conventional Adjuvant TMZ | Dose-dense Adjuvant TMZ
Number analyzed (Participants) | 376 | 384
months
  Unmethylated MGMT: number analyzed (Participants) | 254 | 262
  Unmethylated MGMT | 14.6 [13.2 to 16.5] | 13.3 [12.3 to 14.3]
  Methylated MGMT: number analyzed (Participants) | 122 | 122
  Methylated MGMT | 21.4 [17.6 to 29.0] | 20.2 [15.4 to 25.1]
Statistical Analysis 1: Comparison: Conventional Adjuvant TMZ vs Dose-dense Adjuvant TMZ; Unmethylated MGMT; Test type: Superiority; p = 0.44, Log Rank — One-sided significance level = 0.05; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.82 to 1.19] — Reference level = Conventional adjuvant TMZ
Statistical Analysis 2: Comparison: Conventional Adjuvant TMZ vs Dose-dense Adjuvant TMZ; Methylated MGMT; Test type: Superiority; p = 0.86, Log Rank — One-sided significance level = 0.05; Hazard Ratio (HR) = 1.19, 95% CI 2-sided [0.87 to 1.62] — Reference level = Conventional adjuvant TMZ

4. Secondary Outcome: Median Progression-free Survival Time by MGMT Status
Description: Progression is defined as greater than 25% increase in tumor area (two diameters) provided that the patient has not had his/her dose of steroids decreased since the last evaluation period. Progression-free survival time is defined as time from registration to the date of first progression, death, or last known follow-up (censored). Progression-free survival rates are estimated using the Kaplan-Meier method. A concomitant decrease in steroid dose will rule out a progression designation during the first 2 months after completion of radiation therapy. Tumor tissue submitted at baseline was analyzed to determine MGMT (O[6]-methylguanine-DNA methyltransferase) promoter methylation status (methylated / unmethylated). Analysis occurred after 647 deaths were reported.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 4.4 years.
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Conventional Adjuvant TMZ | Dose-dense Adjuvant TMZ
Number analyzed (Participants) | 376 | 384
months
  Unmethylated MGMT: number analyzed (Participants) | 254 | 262
  Unmethylated MGMT | 5.1 [4.3 to 5.7] | 6.0 [5.5 to 6.5]
  Methylated MGMT: number analyzed (Participants) | 122 | 122
  Methylated MGMT | 6.5 [4.1 to 9.6] | 10.1 [7.9 to 12.4]
Statistical Analysis 1: Comparison: Conventional Adjuvant TMZ vs Dose-dense Adjuvant TMZ; Unmethylated MGMT; Test type: Superiority; p = 0.15, Log Rank — One-sided significance level = 0.05; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.73 to 1.05] — Reference level = Conventional adjuvant TMZ
Statistical Analysis 2: Comparison: Conventional Adjuvant TMZ vs Dose-dense Adjuvant TMZ; Methylated MGMT; Test type: Superiority; p = 0.33, Log Rank — One-sided significance level = 0.05; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.66 to 1.15] — Reference level = Conventional adjuvant TMZ

5. Secondary Outcome: Best Treatment Response by MGMT Status
Description: Response assessed using Response Evaluation Criteria in Solid Tumors (RECIST v1.0): Complete Response (CR), imaging no longer shows enhancing tumor, confirmed by a second scan ≥ 4 weeks later; Partial Response (PR), >=50% decrease in tumor area (two diameters) with patient off all steroids, or on adrenal maintenance only; Minor Response (MR), < 50% decrease in tumor area with patient off all steroids, or on adrenal maintenance only; Stable Disease (SD): scan shows no change with patient receiving stable/decreasing doses of steroids; Progression (P): > 25% increase in tumor area with no decrease in steroid dose since last evaluation. Tumor tissue submitted at baseline was analyzed to determine MGMT (O[6]-methylguanine-DNA methyltransferase) promoter methylation status (methylated / unmethylated). Analysis occurred after 647 deaths were reported.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 4.4 years.
Population: Per the protocol, both arms are combined to compare between MGMT status. MGMT status and treatment response was not available for all randomized eligible participants. Therefore, data was only available for 748/831 randomized eligible patients (arms combined).
Measure: Count of Participants; unit: Participants
Groups:
- Methylated: Methylated MGMT (O[6]-methylguanine-DNA methyltransferase)
- Unmethylated: Unmethylated MGMT (O[6]-methylguanine-DNA methyltransferase)
Arm/Group | Methylated | Unmethylated
Number analyzed (Participants) | 240 | 508
Participants
  Complete Response | 47 | 67
  Partial Response | 34 | 66
  Minor Response | 31 | 55
  Stable Response | 110 | 243
  Progressive Disease | 18 | 77
Statistical Analysis 1: Comparison: Methylated vs Unmethylated; Test type: Superiority; p = 0.012, Chi-squared — Two-sided significance level of 0.05

6. Secondary Outcome: Distribution of Highest Grade AE Reported as Possibly/Probably/Definitely Related to Protocol Treatment
Description: Highest grade adverse event (AE) per subject was counted. Adverse events were graded using the Common Terminology Criteria for Adverse Events (CTCAE) v3.0. Grade refers to the severity of the AE. The CTCAE v3.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild, Grade 2 Moderate, Grade 3 Severe, Grade 4 Life-threatening or disabling, Grade 5 Death related to AE. Analysis occurred after 647 deaths were reported.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 4.4 years.
Population: Randomized eligible patients with any adverse events reported as possibly/probably/definitely related to protocol treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Adjuvant TMZ | Dose-dense Adjuvant TMZ
Number analyzed (Participants) | 351 | 369
Participants
  Grade 0,1,2 | 231 | 175
  Grade 3,4,5 | 120 | 194
Statistical Analysis 1: Comparison: Conventional Adjuvant TMZ vs Dose-dense Adjuvant TMZ; Test type: Superiority; p < 0.001, Chi-squared; Two-sided significance level of 0.05

7. Secondary Outcome: Overall Survival Status by Progression Status at 6 Months
Description: Overall survival time is defined as time from registration to the date of death from any cause or last known follow-up (censored). Overall survival rates are estimated by the Kaplan-Meier method. Progression is defined as greater than 25% increase in tumor area (two diameters) provided that the patient has not had his/her dose of steroids decreased since the last evaluation period.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 4.4 years.
Population: Per the protocol, both arms are combined to compare between 6-month progression status. Eligible pre-randomization participants with any follow-up data.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | No Progression at 6 Months | Progression at 6 Months
Number analyzed (Participants) | 676 | 444
months | 20.7 [19.5 to 22.2] | 10.1 [8.8 to 10.9]
Statistical Analysis 1: Comparison: No Progression at 6 Months vs Progression at 6 Months; Test type: Superiority; p < 0.001, Log Rank — Two-sided test

8. Secondary Outcome: Mean MD Anderson Symptom Inventory Brain Tumor (MDASI-BT) Symptom Severity Score at Cycle 10 for Participants Without Progression After 6 Months of Adjuvant Therapy
Description: The MDASI-BT is a 28-item patient-reported outcome measure assessing symptom severity and resulting interference with daily living in brain cancer patients. All items range from 0 (not present) to 10 (as bad as you can imagine). The symptom severity score is the average of the symptom severity items, given a specified minimum numbers were completed.
Time Frame: Baseline and cycle 10 (approximately 46 weeks)
Population: Cycle 10 questionnaires were not completed by all quality of life (QOL) population participants progression-free at 6 months. Therefore, only 24/96 on the conventional arm and 20/95 on the dose-dense arm had data.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Conventional Adjuvant TMZ: Concurrent radiation therapy with concurrent temozolomide (75 mg/m2) up to 49 doses. Starting four weeks after completion of RT, 100mg/m2 adjuvant temozolomide days 1 to 5 of 28 day cycle for 6 cycles, up to 12 cycles.
- Dose-dense Adjuvant TMZ: Concurrent radiation therapy (RT) with concurrent temozolomide (75 mg/m2) up to 49 doses. Starting four weeks after completion of RT, 75mg/m2 adjuvant temozolomide days 1-21 of 28 day cycle for 6 cycles, up to 12 cycles.
Arm/Group | Conventional Adjuvant TMZ | Dose-dense Adjuvant TMZ
Number analyzed (Participants) | 24 | 20
score on a scale | 1.17 [0.72 to 1.61] | 1.18 [0.68 to 1.69]
Statistical Analysis 1: Comparison: Conventional Adjuvant TMZ vs Dose-dense Adjuvant TMZ; Test type: Superiority; p = 0.96, t-test, 2 sided

9. Secondary Outcome: Mean Neurocognitive Function (NCF) Composite Score at Cycle 10 for Participants Without Progression After 6 Months of Adjuvant Therapy
Description: The NCF Composite score is the arithmetic mean of the Hopkins Verbal Learning Test - Revised (HVLT-R) (Free Recall, Delayed Recall, Delayed Recognition), Trail Making Test Part A (TMTA), Trail Making Test Part B (TMTB), and Controlled Oral Word Association (COWA) test scores, all of which are standardized, adjusting for age, education, and gender as necessary, such that mean is 0 and standard deviation is 1. A participant must have at least 5 of the 6 scores. A higher composite score indicates better neurocognitive function.
Time Frame: Baseline and cycle 10 (approximately 46 weeks)
Population: Cycle 10 questionnaires were not completed by all QOL population participants progression-free at 6 months. Therefore, only 17/96 on the conventional arm and 20/95 on the dose-dense arm had data.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Conventional Adjuvant TMZ | Dose-dense Adjuvant TMZ
Number analyzed (Participants) | 17 | 20
score on a scale | -0.95 [-2.12 to 0.21] | -1.19 [-2.03 to -0.33]
Statistical Analysis 1: Comparison: Conventional Adjuvant TMZ vs Dose-dense Adjuvant TMZ; Test type: Superiority; p = 0.73, t-test, 2 sided

10. Secondary Outcome: Mean EORTC QLQ-C30 Global Health Status Score at Cycle 10 for Participants Without Progression After 6 Months of Adjuvant Therapy
Description: Global Health Status is calculated from two questions on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire [EORTC QLQ]-C30. The question responses range from 1 "very poor" to 7 "excellent" such that a higher response indicates better quality of life (QOL). The mean of these responses is linearly transformed to a range of 0 (worst) to 100 (best).
Time Frame: Baseline and cycle 10 (approximately 46 weeks)
Population: Cycle 10 questionnaires were not completed by all QOL population participants progression-free at 6 months. Therefore, only 24/96 on the conventional arm and 22/95 on the dose-dense arm had data.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Conventional Adjuvant TMZ | Dose-dense Adjuvant TMZ
Number analyzed (Participants) | 24 | 22
score on a scale | 73.3 [64.6 to 81.9] | 69.7 [60.1 to 79.3]
Statistical Analysis 1: Comparison: Conventional Adjuvant TMZ; Test type: Superiority; p = 0.57, t-test, 2 sided

11. Secondary Outcome: Mean Change From Baseline in MD Anderson Symptom Inventory Brain Tumor (MDASI-BT) Symptom Severity Score at Mid-cyle for Cycle 1
Description: The MDASI-BT is a 28-item patient-reported outcome measure assessing symptom severity and resulting interference with daily living in brain cancer patients. All items range from 0 (not present) to 10 (as bad as you can imagine). The symptom severity score is the average of the symptom severity items, given a specified minimum numbers were completed. A score worse than baseline by at least one is considered deterioration. Change is calculated as time point - baseline such that a positive change value indicates worse symptoms compared to baseline.
Time Frame: Baseline and mid-cycle 1 (approximately 12 weeks)
Population: Questionnaires were not completed by all QOL population participants. Therefore, only 41/96 on the conventional arm and 35/95 on the dose-dense arm have both baseline and mid-cycle 1 data.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Conventional Adjuvant TMZ | Dose-dense Adjuvant TMZ
Number analyzed (Participants) | 41 | 35
score on a scale | 0.48 [0.06 to 0.90] | 0.39 [-0.08 to 0.87]
Statistical Analysis 1: Comparison: Conventional Adjuvant TMZ vs Dose-dense Adjuvant TMZ; Test type: Superiority; p = 0.78, t-test, 2 sided

12. Secondary Outcome: Mean Change From Baseline in MD Anderson Symptom Inventory Brain Tumor (MDASI-BT) Symptom Severity Score at Mid-cyle for Cycle 4
Description: as for outcome 11
Time Frame: Baseline and mid-cycle 4 (approximately 24 weeks)
Population: Questionnaires were not completed by all QOL population participants. Therefore, only 32/96 on the conventional arm and 24/95 on the dose-dense arm have both baseline and mid-cycle 4 data.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Conventional Adjuvant TMZ | Dose-dense Adjuvant TMZ
Number analyzed (Participants) | 32 | 24
score on a scale | -0.23 [-0.69 to 0.23] | 0.19 [-0.40 to 0.77]
Statistical Analysis 1: Comparison: Conventional Adjuvant TMZ vs Dose-dense Adjuvant TMZ; Test type: Superiority; p = 0.24, t-test, 2 sided

13. Secondary Outcome: Mean Change From Baseline in EORTC QLQ-C30 Global Health Status Score at Mid-cyle for Cycle 1
Description: Global Health Status is calculated from two questions on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire [EORTC QLQ]-C30. The question responses range from 1 "very poor" to 7 "excellent" such that a higher response indicates better quality of life (QOL). The mean of these responses is linearly transformed to a range of 0 (worst) to 100 (best). Change is calculated as time point - baseline such that a positive change value indicates worse symptoms compared to baseline.
Time Frame: Baseline and mid-cycle 1 (approximately 12 weeks)
Population: Questionnaires were not completed by all QOL population participants. Therefore, only 40/96 on the conventional arm and 38/95 on the dose-dense arm have both baseline and mid-cycle 1 data.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Conventional Adjuvant TMZ | Dose-dense Adjuvant TMZ
Number analyzed (Participants) | 40 | 38
score on a scale | -4.58 [-12.63 to 3.47] | -2.63 [-11.37 to 6.10]
Statistical Analysis 1: Comparison: Conventional Adjuvant TMZ vs Dose-dense Adjuvant TMZ; Test type: Superiority; p = 0.74, t-test, 2 sided

14. Secondary Outcome: Mean Change From Baseline in EORTC QLQ-C30 Global Health Status Score at Mid-cyle for Cycle 4
Description: as for outcome 13
Time Frame: Baseline and mid-cycle 4 (approximately 24 weeks)
Population: Questionnaires were not completed by all QOL population participants. Therefore, only 30/96 on the conventional arm and 23/95 on the dose-dense arm have both baseline and mid-cycle 4 data.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Conventional Adjuvant TMZ | Dose-dense Adjuvant TMZ
Number analyzed (Participants) | 30 | 23
score on a scale | -2.78 [-13.87 to 8.32] | -0.72 [-11.91 to 10.46]
Statistical Analysis 1: Comparison: Conventional Adjuvant TMZ vs Dose-dense Adjuvant TMZ; Test type: Superiority; p = 0.79, t-test, 2 sided

15. Secondary Outcome: Change From Baseline in Mean EORTC QLQ-C30 Global Health Status
Description: Global Health Status is calculated from two questions on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire [EORTC QLQ]-C30. The question responses range from 1 "very poor" to 7 "excellent" such that a higher response indicates better quality of life (QOL). The mean of these responses is linearly transformed to a range of 0 (worst) to 100 (best). Change from baseline was calculated as time point value - baseline value with a positive change value indicating improved QOL from baseline.
Time Frame: Baseline, 10,12, 22, 24, and 46 weeks
Population: Questionnaires were not completed by all QOL population participants. Therefore, the number of participants reported below are the number with the relevant questions answered at baseline and the given time point on each arm.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Conventional Adjuvant TMZ | Dose-dense Adjuvant TMZ
Number analyzed (Participants) | 96 | 95
score on a scale
  Week 10 (Cycle 1): number analyzed (Participants) | 70 | 72
  Week 10 (Cycle 1) | 0.0 [-6.1 to 6.1] | -2.9 [-8.7 to 2.9]
  Week 12 (Cycle 1.5): number analyzed (Participants) | 40 | 38
  Week 12 (Cycle 1.5) | -4.6 [-12.6 to 3.5] | -2.7 [-11.3 to 6.1]
  Week 22 (Cycle 4): number analyzed (Participants) | 48 | 38
  Week 22 (Cycle 4) | 3.9 [-2.5 to 10.4] | -4.4 [-12.1 to 3.3]
  Week 24 (Cycle 4.5): number analyzed (Participants) | 30 | 23
  Week 24 (Cycle 4.5) | -2.8 [-13.9 to 8.3] | -0.7 [-11.9 to 10.5]
  Week 46 (Cycle 10): number analyzed (Participants) | 23 | 22
  Week 46 (Cycle 10) | 5.4 [-7.5 to 18.3] | -1.9 [-9.8 to 6.0]
Statistical Analysis 1: Comparison: Conventional Adjuvant TMZ vs Dose-dense Adjuvant TMZ; A mixed effects model was run with EORTC QLQ-C30 Global Health Status Score (baseline, 10,12, 22, 24, and 46 weeks) as the outcome of interest. Treatment arm, recursive partitioning analysis (RPA) class, MGMT status, and time were included in the model. Treatment arm is reported here; Test type: Superiority; p = 0.2184, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept effects are not shown.)
Statistical Analysis 2: Comparison: Conventional Adjuvant TMZ vs Dose-dense Adjuvant TMZ; A mixed effects model was run with EORTC QLQ-C30 Global Health Status Score (baseline, 10,12, 22, 24, and 46 weeks) as the outcome of interest. Treatment arm, RPA class, MGMT status, and time were included in the model. RPA class is reported here; Test type: Superiority; p = 0.0763, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept effects are not shown.)
Statistical Analysis 3: Comparison: Conventional Adjuvant TMZ vs Dose-dense Adjuvant TMZ; A mixed effects model was run with EORTC QLQ-C30 Global Health Status Score (baseline, 10,12, 22, 24, and 46 weeks) as the outcome of interest. Treatment arm, RPA class, MGMT status, and time were included in the model. MGMT status is reported here; Test type: Superiority; p = 0.5235, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept effects are not shown.)

16. Secondary Outcome: Number of Participants With Deterioration From Baseline in MD Anderson Symptom Inventory Brain Tumor (MDASI-BT) Symptom Severity Score at Cycle 4
Description: The MDASI-BT is a 28-item patient-reported outcome measure assessing symptom severity and resulting interference with daily living in brain cancer patients. All items range from 0 (not present) to 10 (as bad as you can imagine). The symptom severity score is the average of the symptom severity items, given a specified minimum numbers were completed. A score worse than baseline by at least one is considered deterioration.
Time Frame: baseline and cycle 4 (approximately 22 weeks)
Population: Questionnaires were not completed by all QOL population participants. Therefore, only 51/96 on the conventional arm and 40/95 on the dose-dense arm have both baseline and cycle 4 data
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Adjuvant TMZ | Dose-dense Adjuvant TMZ
Number analyzed (Participants) | 51 | 40
Participants | 5 | 11
Statistical Analysis 1: Comparison: Conventional Adjuvant TMZ vs Dose-dense Adjuvant TMZ; Test type: Superiority; p = 0.03, Z-test of two proportions

17. Secondary Outcome: Number of Participants With Deterioration From Baseline in MD Anderson Symptom Inventory Brain Tumor (MDASI-BT) Interference Score at Cycle 4
Description: The MDASI-BT is a 28-item patient-reported outcome measure assessing symptom severity and resulting interference with daily living in brain cancer patients. All items range from 0 (did not interfere) to 10 (interfered completely). The symptom interference score is the average of the symptom interference items, given a specified minimum numbers were completed. A score worse than baseline by at least one is considered deterioration.
Time Frame: baseline and cycle 4 (approximately 22 weeks)
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Adjuvant TMZ | Dose-dense Adjuvant TMZ
Number analyzed (Participants) | 51 | 40
Participants | 7 | 13
Statistical Analysis 1: Comparison: Conventional Adjuvant TMZ vs Dose-dense Adjuvant TMZ; Test type: Superiority; p = 0.03, Z-test of two proportions

18. Secondary Outcome: Number of Participants With Deterioration From Baseline in MD Anderson Symptom Inventory Brain Tumor (MDASI-BT) Symptom Severity Score and EORTC QLQ-C30 Global Health Status Score (GHS) at Cycle 1
Description: * The MDASI-BT is a 28-item patient-reported outcome measure assessing symptom severity (SS) and resulting interference with daily living in brain cancer patients. All items range from 0 (not present) to 10 (as bad as you can imagine). A SS score is the average of the SS items, given a specified minimum numbers were completed. A score worse than baseline by at least one is considered deterioration.
  * Global Health Status is calculated from two questions on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire [EORTC QLQ]-C30. The question responses range from 1 (very poor) to 7 (excellent) such that a higher response indicates better quality of life (QOL). The mean of these responses is linearly transformed to a range of 0 (worst) to 100 (best). A score worse than baseline by at least 10 is considered deterioration.
  * The 2x2 frequency table of SS deterioration vs. GHS deterioration is presented as four rows.
Time Frame: baseline and cycle 1 (approximately 10 weeks)
Population: Per the protocol, both arms are combined. Questionnaires were not completed by all QOL population participants. Therefore, only 136/191 have both MDASI-BT and EORTC QLQ-C30 at baseline and cycle 1.
Measure: Count of Participants; unit: Participants
Groups:
- Both Arms Combined: Concurrent radiation therapy with concurrent temozolomide (75 mg/m2) up to 49 doses. Starting four weeks after completion of RT, either [100mg/m2 adjuvant temozolomide days 1 to 5 of 28 day cycle] or [75mg/m2 adjuvant temozolomide days 1-21 of 28 day cycle] for 6 cycles, up to 12 cycles.
Arm/Group | Both Arms Combined
Number analyzed (Participants) | 136
Participants
  Symptom Severity and GHS deterioration | 18
  Symptom Severity deterioration only | 9
  GHS deterioratoin only | 31
  No deterioration | 78
Statistical Analysis 1: Comparison: Both Arms Combined; Test type: Superiority; p = 0.0002, Chi-squared; Two-sided test

19. Secondary Outcome: Number of Participants With Deterioration From Baseline in MD Anderson Symptom Inventory Brain Tumor (MDASI-BT) Symptom Severity Score and EORTC QLQ-C30 Global Health Status Score (GHS) at Cycle 4
Description: as for outcome 18
Time Frame: baseline and cycle 4 (approximately 22 weeks)
Population: Both arms are combined per the protocol. Questionnaires were not completed by all QOL population participants. Therefore, only 86/191 have both MDASI-BT and EORTC QLQ-C30 at baseline and cycle 4.
Measure: Count of Participants; unit: Participants
Arm/Group | Both Arms Combined
Number analyzed (Participants) | 86
Participants
  Symptom Severity and GHS deterioration | 10
  Symptom Severity deterioration only | 5
  GHS deterioration Only | 18
  No deterioration | 53
Statistical Analysis 1: Comparison: Both Arms Combined; Test type: Superiority; p = 0.005, Fisher Exact; Two-sided test

20. Secondary Outcome: Number of Participants With Deterioration From Baseline in MD Anderson Symptom Inventory Brain Tumor (MDASI-BT) Symptom Severity Score and EORTC QLQ-C30 Global Health Status Score (GHS) at Cycle 10
Description: as for outcome 18
Time Frame: baseline and cycle 10 (approximately 46 weeks)
Population: Both arms are combined per the protocol. Questionnaires were not completed by all QOL population participants. Therefore, only 44/191 have both MDASI-BT and EORTC QLQ-C30 at baseline and cycle 10.
Measure: Count of Participants; unit: Participants
Arm/Group | Both Arms Combined
Number analyzed (Participants) | 44
Participants
  Symptom Severity and GHS deterioration | 5
  Symptom Severity deterioration only | 4
  GHS deterioration only | 5
  No deterioration | 30
Statistical Analysis 1: Comparison: Both Arms Combined; Test type: Superiority; p = 0.018, Fisher Exact; Two-sided test

21. Secondary Outcome: Mean MD Anderson Symptom Inventory Brain Tumor (MDASI-BT) Symptom Severity Score Over Time
Description: as for outcome 8
Time Frame: Baseline, 10, 12, 22, 24, and 46 weeks
Population: as for outcome 15
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Conventional Adjuvant TMZ | Dose-dense Adjuvant TMZ
Number analyzed (Participants) | 95 | 96
score on a scale
  Baseline: number analyzed (Participants) | 88 | 86
  Baseline | 1.3 [1.0 to 1.5] | 1.1 [0.8 to 1.4]
  Week 10 (Cycle 1): number analyzed (Participants) | 73 | 74
  Week 10 (Cycle 1) | 1.4 [1.1 to 1.7] | 1.4 [1.1 to 1.6]
  Week 12 (Cycle 1.5): number analyzed (Participants) | 41 | 37
  Week 12 (Cycle 1.5) | 1.6 [1.2 to 2.1] | 1.5 [1.1 to 1.8]
  Week 22 (Cycle 4): number analyzed (Participants) | 51 | 40
  Week 22 (Cycle 4) | 1.0 [0.7 to 1.3] | 1.2 [0.9 to 1.5]
  Week 24 (Cycle 4.5): number analyzed (Participants) | 32 | 24
  Week 24 (Cycle 4.5) | 1.0 [0.7 to 1.3] | 1.1 [0.7 to 1.6]
  Week 46 (Cycle 10): number analyzed (Participants) | 24 | 22
  Week 46 (Cycle 10) | 1.2 [0.7 to 1.6] | 1.1 [0.7 to 1.6]
Statistical Analysis 1: Comparison: Conventional Adjuvant TMZ vs Dose-dense Adjuvant TMZ; A mixed effects model was run with MDASI Symptom Severity Score (baseline, 10, 12, 22, 24, 46 weeks) as the outcome of interest. Treatment arm, recursive partitioning analysis (RPA) class, MGMT status, and time were included in the model. Treatment arm is reported here; Test type: Superiority — Each explanatory variable is reported separately. (Time and intercept effects are not shown.); p = 0.1702, Mixed Models Analysis
Statistical Analysis 2: Comparison: Conventional Adjuvant TMZ vs Dose-dense Adjuvant TMZ; A mixed effects model was run with EORTC QLQ-C30 Global Health Status Score (baseline, 10, 12, 22, 24, 46 weeks) as the outcome of interest. Treatment arm, recursive partitioning analysis (RPA) class, MGMT status, and time were included in the model. RPA is reported here; Test type: Superiority; p = 0.8159, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept effects are not shown.)
Statistical Analysis 3: Comparison: Conventional Adjuvant TMZ vs Dose-dense Adjuvant TMZ; A mixed effects model was run with EORTC QLQ-C30 Global Health Status Score (baseline, 10, 12, 22, 24, 46 weeks) as the outcome of interest. Treatment arm, recursive partitioning analysis (RPA) class, MGMT status, and time were included in the model. MGMT status is reported here; Test type: Superiority; p = 0.2174, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept effects are not shown.)

22. Secondary Outcome: Determination of Impactful Baseline Instruments on Overall Survival
Description: Overall survival time is defined as time from registration/randomization to the date of death from any cause or last known follow-up (censored). Overall survival rates are estimated by the Kaplan-Meier method. The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire [EORTC QLQ]-C30 subscales are calculated as the mean of component items, then standardized such that subscale scores range from 0 to 100. A high score for a functional scale represents a healthy level of functioning. Controlled Oral Word Association (COWA) score is the sum of correct responses with a range of 0 to infinity. A higher score indicates better functioning. Hopkins Verbal Learning Test - Revised (HVLT-R) score ranges from 0 to 36 for total recall is 0 to 36, 0 to 12 for delayed recall, and -12 to 12 for recognition. A higher score indicates better functioning.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 4.4 years.
Population: Both arms are combined per the protocol. Questionnaires/assessments were not completed by all QOL population participants. Therefore, only 154/191 have COWA, EORTC QLQ-C30, and HVLT-R baseline assessments (final model covariates)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Both Arms Combined
Number analyzed (Participants) | 154
months | 17.5 [14.0 to 20.9]
Statistical Analysis 1: Comparison: Both Arms Combined; A Cox proportional hazards model was run with overall survival as the outcome of interest and baseline scores as continuous covariates. The final model was determined from stepwise selection. EORTC physical functioning, EORTC role functioning, standardized HVLT-R recognition, standardized HVLT-R recall, and standardized COWA were included in the initial model. EORTC physical functioning is reported here; Test type: Other; p = 0.023, Regression, Cox
Statistical Analysis 2: Comparison: Both Arms Combined; A Cox proportional hazards model was run with overall survival as the outcome of interest and baseline scores as continuous covariates. The final model was determined from stepwise selection. EORTC physical functioning, EORTC role functioning, standardized HVLT-R recognition, standardized HVLT-R recall, and standardized COWA were included in the initial model. Standardized HVLT-R recognition is reported here; Test type: Other; p = 0.043, Regression, Cox
Statistical Analysis 3: Comparison: Both Arms Combined; A Cox proportional hazards model was run with overall survival as the outcome of interest and baseline scores as continuous covariates. The final model was determined from stepwise selection. EORTC physical functioning, EORTC role functioning, standardized HVLT-R recognition, standardized HVLT-R recall, and standardized COWA were included in the initial model. Standardized COWA is reported here; Test type: Other; p = 0.021, Regression, Cox

23. Secondary Outcome: Mean Neurocognitive Function (NCF) Composite Score Over Time
Description: The NCF Composite score is the arithmetic mean of the HVLT-R (Free Recall, Delayed Recall, Delayed Recognition), TMTA, TMTB, and COWA scores, all of which are standardized, adjusting for age, education, and gender as necessary, such that mean is 0 and standard deviation is 1. A participant must have at least 5 of the 6 scores. A higher composite score indicates better neurocognitive function.
Time Frame: Baseline, 10, 22, and 46 weeks
Population: Questionnaires were not completed by all QOL population participants. Therefore, the number of participants reported below are the number with data at baseline and the given time point on each arm.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Conventional Adjuvant TMZ | Dose-dense Adjuvant TMZ
Number analyzed (Participants) | 96 | 95
score on a scale
  Baseline: number analyzed (Participants) | 80 | 85
  Baseline | -1.2 [-1.6 to -0.9] | -1.5 [-1.8 to -1.1]
  Week 10 (Cycle 1): number analyzed (Participants) | 67 | 63
  Week 10 (Cycle 1) | -1.3 [-1.7 to -1.0] | -1.45 [-1.9 to -1.0]
  Week 22 (Cycle 4): number analyzed (Participants) | 39 | 35
  Week 22 (Cycle 4) | -1.1 [-1.6 to -0.6] | -1.3 [-2.0 to -0.6]
  Week 46 (Cycle 10): number analyzed (Participants) | 17 | 20
  Week 46 (Cycle 10) | -1.0 [-2.1 to 0.2] | -1.2 [-2.0 to -0.3]
Statistical Analysis 1: Comparison: Conventional Adjuvant TMZ vs Dose-dense Adjuvant TMZ; A mixed effects model was run with NCF Composite Score (baseline, 10, 22, 46 weeks) as the outcome of interest. Treatment arm, recursive partitioning analysis (RPA) class, MGMT status, and time were included in the model. Treatment arm is reported here; Test type: Superiority; p = 0.2357, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept effects are not shown.)
Statistical Analysis 2: Comparison: Conventional Adjuvant TMZ vs Dose-dense Adjuvant TMZ; A mixed effects model was run with NCF Composite Score (baseline, 10, 22, 46 weeks) as the outcome of interest. Treatment arm, recursive partitioning analysis (RPA) class, MGMT status, and time were included in the model. RPA is reported here; Test type: Superiority; p = 0.0147, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept effects are not shown.)
Statistical Analysis 3: Comparison: Conventional Adjuvant TMZ vs Dose-dense Adjuvant TMZ; A mixed effects model was run with NCF Composite Score (baseline, 10, 22, 46 weeks) as the outcome of interest. Treatment arm, recursive partitioning analysis (RPA) class, MGMT status, and time were included in the model. MGMT Status is reported here; Test type: Superiority; p = 0.457, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept effects are not shown.)

24. Secondary Outcome: Number of Participants With Deterioration From Baseline in MD Anderson Symptom Inventory Brain Tumor (MDASI-BT) Cognitive Score and Hopkins Verbal Learning Test - Revised (HVLT-R) Delayed Recognition Score at Cycle 1
Description: * The MDASI-BT is a 28-item patient-reported outcome measure assessing symptom severity (SS) and resulting interference with daily living in brain cancer patients. All items range from 0 (not present) to 10 (as bad as you can imagine). A SS score is the average of the SS items, given a specified minimum numbers were completed. A score worse than baseline by at least one is considered deterioration.
  * The HVLT-R Delayed Recognition raw score is the number of of correctly identified words minus the number of incorrectly identified words from a list of words including 12 nouns memorized 20 minutes prior. The raw score ranges from -12 to 12. with a higher score indicates better functioning. Scores are standardized (mean 0, standard deviation 1), adjusting for age,education, and gender as necessary. A score worse than baseline by at least two is considered deterioration.
  * The 2x2 frequency table of SS deterioration vs. HVLT-R deterioration is presented as four rows.
Time Frame: baseline and cycle 1 (approximately 10 weeks)
Population: Both arms are combined per the protocol. Questionnaires/assessments were not completed by all QOL population participants. Therefore, only 116/191 have both MDASI-BT and HVLT-R at baseline and cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Both Arms Combined
Number analyzed (Participants) | 116
Participants
  Cognitive and HVLT-R deterioration | 10
  Cognitive deterioration only | 12
  HVLT-R deterioration only | 20
  No deterioration | 74
Statistical Analysis 1: Comparison: Both Arms Combined; Test type: Superiority; p = 0.02, Chi-squared; Two-sided test

25. Secondary Outcome: Number of Participants With Deterioration From Baseline in MD Anderson Symptom Inventory Brain Tumor (MDASI-BT) Cognitive Score and Hopkins Verbal Learning Test - Revised (HVLT-R) Delayed Recognition (DR) Score at Cycle 4
Description: as for outcome 24
Time Frame: baseline and cycle 4 (approximately 22 weeks)
Population: Both arms are combined per the protocol. Questionnaires/assessments were not completed by all QOL population participants. Therefore, only 71/191 have both MDASI-BT and HVLT-R at baseline and cycle 4.
Measure: Count of Participants; unit: Participants
Arm/Group | Both Arms Combined
Number analyzed (Participants) | 71
Participants
  Cognitive and Delayed Recognition deterioration | 3
  Cognitive deterioration only | 9
  Delayed Recognition deterioration only | 14
  No deterioration | 45
Statistical Analysis 1: Comparison: Both Arms Combined; Test type: Superiority; p = 0.99, Fisher Exact; Two-sided test

26. Secondary Outcome: Number of Participants With Deterioration From Baseline in MD Anderson Symptom Inventory Brain Tumor (MDASI-BT) Cognitive Score and Hopkins Verbal Learning Test - Revised (HVLT-R) Delayed Recognition (DR) Score at Cycle 10
Description: as for outcome 24
Time Frame: baseline and cycle 10 (approximately 46 weeks)
Population: Both arms are combined per the protocol. Questionnaires/assessments were not completed by all QOL population participants. Therefore, only 36/191 have both MDASI-BT and HVLT-R at baseline and cycle 10.
Measure: Count of Participants; unit: Participants
Arm/Group | Both Arms Combined
Number analyzed (Participants) | 36
Participants
  Cognitive and Delayed Recognition deterioration | 3
  Cognitive deterioration only | 6
  Delayed Recognition deterioration only | 4
  No deterioration | 23
Statistical Analysis 1: Comparison: Both Arms Combined; Test type: Superiority; p = 0.33, Fisher Exact; Two-sided test

ADVERSE EVENTS:
Description: Eligible participants with adverse event data: concurrent RT and TMZ only arm (not randomized): 285/292; conventional adjuvant TMZ arm: 409/411; dose-dense adjuvant TMZ arm: 420/422.
Groups:
- No Adjuvant TMZ (Not Randomized): Concurrent radiation therapy (RT) with concurrent temozolomide (75 mg/m2) up to 49 doses. Not randomized to either adjuvant TMZ arm.
Arm/Group | No Adjuvant TMZ (Not Randomized) | Conventional Adjuvant TMZ | Dose-dense Adjuvant TMZ
Serious Adverse Events (participants affected / at risk) | 105/285 | 131/409 | 142/420
Other Adverse Events (participants affected / at risk) | 216/285 | 376/409 | 392/420
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | No Adjuvant TMZ (Not Randomized) (N=285) | Conventional Adjuvant TMZ (N=409) | Dose-dense Adjuvant TMZ (N=420)
Blood/bone marrow - Other: (Blood and lymphatic system disorders) | 0 | 2 | 1
Bone marrow depression NOS (Blood and lymphatic system disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 1
Haemolysis NOS (Blood and lymphatic system disorders) | 1 | 0 | 1
Hemoglobin (Blood and lymphatic system disorders) | 12 | 6 | 5
Thrombotic microangiopathy NOS (Blood and lymphatic system disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 3 | 2
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 1
Cardiac General - Other: (Cardiac disorders) | 2 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 2
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1
Cushingoid (Endocrine disorders) | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 1
Extraocular muscle disorder (Eye disorders) | 0 | 2 | 0
Ocular/visual - Other: (Eye disorders) | 0 | 2 | 0
Photopsia (Eye disorders) | 1 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1
Abdominal pain NOS (Gastrointestinal disorders) | 0 | 3 | 2
Colitis NOS (Gastrointestinal disorders) | 2 | 1 | 0
Colonic perforation (Gastrointestinal disorders) | 1 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 4 | 0
Diarrhoea NOS (Gastrointestinal disorders) | 1 | 2 | 3
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis NOS (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal - Other: (Gastrointestinal disorders) | 1 | 2 | 1
Nausea (Gastrointestinal disorders) | 6 | 7 | 11
Oseophagitis NOS (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis NOS (Gastrointestinal disorders) | 0 | 1 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal stricture NOS (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting NOS (Gastrointestinal disorders) | 5 | 5 | 9
Chest pain (General disorders) | 1 | 0 | 0
Constitutional Symptoms - Other: (General disorders) | 1 | 0 | 0
Death NOS (General disorders) | 2 | 1 | 0
Disease progression NOS (General disorders) | 6 | 3 | 2
Edema: head and neck: (General disorders) | 0 | 0 | 2
Edema: limb: (General disorders) | 2 | 2 | 0
Fatigue (General disorders) | 9 | 9 | 11
Gait abnormal NOS (General disorders) | 2 | 1 | 0
Influenza-like illness (General disorders) | 0 | 1 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0
Pain - Other: (General disorders) | 1 | 0 | 0
Pain NOS (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 6 | 5 | 7
Rigors (General disorders) | 1 | 1 | 0
Sudden death (General disorders) | 2 | 0 | 1
Cholecystitis NOS (Hepatobiliary disorders) | 0 | 1 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0
Allergy/immunology - Other: (Immune system disorders) | 1 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 1 | 0
Hypersensitivity NOS (Immune system disorders) | 3 | 0 | 3
Abdominal infection (Infections and infestations) | 0 | 1 | 0
Arthritis infective NOS (Infections and infestations) | 0 | 1 | 1
Bladder infection NOS (Infections and infestations) | 0 | 1 | 0
Bone infection NOS (Infections and infestations) | 0 | 1 | 0
Bronchitis NOS (Infections and infestations) | 1 | 0 | 0
Encephalitis NOS (Infections and infestations) | 1 | 0 | 1
Eye infection NOS (Infections and infestations) | 0 | 0 | 1
Infection - Other: (Infections and infestations) | 3 | 4 | 2
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Biliary tree (Infections and infestations) | 0 | 0 | 1
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Bladder (urinary) (Infections and infestations) | 0 | 0 | 1
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Bronchus (Infections and infestations) | 1 | 0 | 0
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Kidney (Infections and infestations) | 0 | 0 | 1
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Lung (pneumonia) (Infections and infestations) | 1 | 2 | 4
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Meninges (meningitis) (Infections and infestations) | 1 | 0 | 0
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Rectum (Infections and infestations) | 0 | 1 | 0
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Soft tissue NOS (Infections and infestations) | 1 | 0 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils: Blood (Infections and infestations) | 1 | 0 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils: Esophagus (Infections and infestations) | 1 | 0 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils: Nerve-peripheral (Infections and infestations) | 0 | 1 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils: Wound (Infections and infestations) | 2 | 2 | 0
Infection with unknown ANC: Lung (pneumonia) (Infections and infestations) | 0 | 1 | 0
Infection with unknown ANC: Meninges (meningitis) (Infections and infestations) | 1 | 0 | 0
Infection with unknown ANC: Skin (cellulitis) (Infections and infestations) | 1 | 1 | 0
Infectous meningitis (Infections and infestations) | 0 | 0 | 1
Opportunisitic infection (Infections and infestations) | 1 | 0 | 5
Pneumonia NOS (Infections and infestations) | 0 | 4 | 3
Respiratory tract infection NOS (Infections and infestations) | 0 | 1 | 0
Rhinitis infective (Infections and infestations) | 0 | 1 | 0
Sepsis NOS (Infections and infestations) | 0 | 0 | 1
Sinusitis NOS (Infections and infestations) | 0 | 0 | 1
Skin infection (Infections and infestations) | 1 | 5 | 1
Urinary tract infection NOS (Infections and infestations) | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 2
Fracture NOS (Injury, poisoning and procedural complications) | 2 | 1 | 3
Vascular access NOS complication (Injury, poisoning and procedural complications) | 2 | 3 | 1
Alanine aminotransferase increased (Investigations) | 5 | 3 | 3
Aspartate aminotransferase increased (Investigations) | 4 | 3 | 2
Blood alkaline phosphatase increased (Investigations) | 2 | 3 | 3
Blood amylase increased (Investigations) | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 4 | 3 | 2
Blood creatinine increased (Investigations) | 2 | 0 | 2
CD4 lymphocytes decreased (Investigations) | 0 | 0 | 6
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0
Inappropriate antidiuretic hormone secretion (Investigations) | 1 | 1 | 0
Leukopenia NOS (Investigations) | 17 | 15 | 14
Lipase increased (Investigations) | 0 | 1 | 1
Lymphopenia (Investigations) | 11 | 5 | 23
Metabolic/laboratory - Other: (Investigations) | 1 | 3 | 1
Neutrophil count (Investigations) | 20 | 15 | 11
Platelet count decreased (Investigations) | 34 | 20 | 16
Prothrombin time prolonged (Investigations) | 1 | 0 | 0
Troponin I increased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 1 | 1
Acidosis NOS (Metabolism and nutrition disorders) | 0 | 1 | 1
Alkalosis NOS (Metabolism and nutrition disorders) | 1 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 2 | 5
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 3 | 7
Hyperglycaemia NOS (Metabolism and nutrition disorders) | 0 | 6 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 2 | 4
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypoglycemia NOS (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 3 | 4 | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 5 | 6 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle weakness NOS (Musculoskeletal and connective tissue disorders) | 2 | 2 | 10
Muscle weakness, generalized or specific area (not due to neuropathy): Extremity-lower (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Muscle weakness, generalized or specific area (not due to neuropathy): Extremity-upper (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle weakness, generalized or specific area (not due to neuropathy): Left-sided (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle weakness, generalized or specific area (not due to neuropathy): Right-sided (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Musculoskeletal/soft tissue - Other: (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Ataxia (Nervous system disorders) | 0 | 0 | 4
CNS necrosis/cystic progression: (Nervous system disorders) | 0 | 2 | 1
Cerebral ischaemia (Nervous system disorders) | 3 | 3 | 4
Cerebrospinal fluid leak (Nervous system disorders) | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1 | 5
Convulsions NOS (Nervous system disorders) | 9 | 23 | 24
Depressed level of consciousness (Nervous system disorders) | 2 | 2 | 3
Diaphragmatic paralysis (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 5 | 3
Dysgeusia (Nervous system disorders) | 0 | 2 | 1
Encephalopathy (Nervous system disorders) | 1 | 1 | 2
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 6 | 9 | 7
Hemorrhagic stroke (Nervous system disorders) | 4 | 0 | 0
Hydrocephalus acquired (Nervous system disorders) | 0 | 3 | 2
Hyperreflexia (Nervous system disorders) | 2 | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 3 | 3
Mental status changes (Nervous system disorders) | 1 | 1 | 1
Muscle weakness, generalized or specific area (not due to neuropathy): Facial (Nervous system disorders) | 0 | 1 | 0
Neuralgia NOS (Nervous system disorders) | 0 | 1 | 0
Neurology - Other: (Nervous system disorders) | 4 | 3 | 4
Neuropathy: cranial: CN VIII Hearing and balance (Nervous system disorders) | 1 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 8 | 7
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1 | 2
Speech disorder (Nervous system disorders) | 1 | 3 | 2
Syncope (Nervous system disorders) | 1 | 1 | 2
Syncope vasovagal (Nervous system disorders) | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 1 | 1
Agitation (Psychiatric disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 5 | 12 | 10
Depression (Psychiatric disorders) | 1 | 4 | 4
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Libido decreased (Psychiatric disorders) | 0 | 0 | 1
Personality change (Psychiatric disorders) | 0 | 3 | 0
Psychosis aggravated (Psychiatric disorders) | 1 | 2 | 0
Cystitis NOS (Renal and urinary disorders) | 0 | 0 | 1
Renal failure NOS (Renal and urinary disorders) | 2 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Erectile dysfunction NOS (Reproductive system and breast disorders) | 0 | 0 | 1
Scrotal pain (Reproductive system and breast disorders) | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 7
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 6
Nasal cavity/paranasal sinus reactions: (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Pneumonitis NOS (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 6
Pulmonary/upper respiratory - Other: (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Respiratory tract hemorrhage NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acne NOS (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermatitis exfoliative NOS (Skin and subcutaneous tissue disorders) | 1 | 1 | 3
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hematoma (Vascular disorders) | 0 | 0 | 2
Hypotension NOS (Vascular disorders) | 3 | 1 | 3
Thrombosis (Vascular disorders) | 15 | 15 | 19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | No Adjuvant TMZ (Not Randomized) (N=285) | Conventional Adjuvant TMZ (N=409) | Dose-dense Adjuvant TMZ (N=420)
Hemoglobin (Blood and lymphatic system disorders) | 69 | 142 | 171
Hearing impaired (Ear and labyrinth disorders) | 8 | 27 | 20
Ocular/visual - Other: (Eye disorders) | 16 | 37 | 27
Vision blurred (Eye disorders) | 19 | 48 | 54
Abdominal pain NOS (Gastrointestinal disorders) | 5 | 17 | 25
Constipation (Gastrointestinal disorders) | 58 | 135 | 129
Diarrhoea NOS (Gastrointestinal disorders) | 12 | 50 | 75
Dry mouth (Gastrointestinal disorders) | 7 | 22 | 26
Dyspepsia (Gastrointestinal disorders) | 11 | 30 | 32
Nausea (Gastrointestinal disorders) | 79 | 226 | 228
Stomatitis (Gastrointestinal disorders) | 9 | 20 | 24
Vomiting NOS (Gastrointestinal disorders) | 32 | 114 | 117
Edema: head and neck: (General disorders) | 7 | 15 | 27
Edema: limb: (General disorders) | 18 | 49 | 54
Fatigue (General disorders) | 134 | 292 | 320
Pain - Other: (General disorders) | 3 | 29 | 23
Pyrexia (General disorders) | 8 | 25 | 27
Dermatitis radiation NOS (Injury, poisoning and procedural complications) | 43 | 97 | 103
Radiation recall syndrome (Injury, poisoning and procedural complications) | 10 | 20 | 26
Alanine aminotransferase increased (Investigations) | 41 | 100 | 109
Aspartate aminotransferase increased (Investigations) | 21 | 64 | 70
Blood alkaline phosphatase increased (Investigations) | 17 | 46 | 49
Blood creatinine increased (Investigations) | 7 | 25 | 32
CD4 lymphocytes decreased (Investigations) | 0 | 13 | 32
Leukopenia NOS (Investigations) | 44 | 152 | 190
Lymphopenia (Investigations) | 49 | 170 | 179
Metabolic/laboratory - Other: (Investigations) | 16 | 39 | 38
Neutrophil count (Investigations) | 18 | 89 | 107
Platelet count decreased (Investigations) | 53 | 161 | 163
Weight decreased (Investigations) | 12 | 54 | 73
Anorexia (Metabolism and nutrition disorders) | 48 | 113 | 140
Hyperglycaemia NOS (Metabolism and nutrition disorders) | 50 | 116 | 130
Hypernatremia (Metabolism and nutrition disorders) | 4 | 21 | 20
Hypoalbuminemia (Metabolism and nutrition disorders) | 20 | 46 | 56
Hypocalcemia (Metabolism and nutrition disorders) | 20 | 39 | 45
Hypoglycemia NOS (Metabolism and nutrition disorders) | 4 | 21 | 22
Hypokalemia (Metabolism and nutrition disorders) | 18 | 46 | 51
Hyponatremia (Metabolism and nutrition disorders) | 22 | 48 | 60
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 27 | 32
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 23 | 23
Muscle weakness NOS (Musculoskeletal and connective tissue disorders) | 19 | 41 | 49
Muscle weakness, generalized or specific area (not due to neuropathy): Extremity-lower (Musculoskeletal and connective tissue disorders) | 11 | 33 | 26
Muscle weakness, generalized or specific area (not due to neuropathy): Left-sided (Musculoskeletal and connective tissue disorders) | 4 | 24 | 16
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 13 | 24
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 22 | 30
Ataxia (Nervous system disorders) | 23 | 56 | 54
Cognitive disorder (Nervous system disorders) | 11 | 31 | 37
Convulsions NOS (Nervous system disorders) | 34 | 80 | 87
Depressed level of consciousness (Nervous system disorders) | 8 | 15 | 23
Dizziness (Nervous system disorders) | 25 | 93 | 75
Dysgeusia (Nervous system disorders) | 19 | 43 | 63
Headache (Nervous system disorders) | 69 | 193 | 199
Hyperreflexia (Nervous system disorders) | 9 | 24 | 23
Memory impairment (Nervous system disorders) | 29 | 84 | 85
Neurology - Other: (Nervous system disorders) | 7 | 34 | 34
Peripheral motor neuropathy (Nervous system disorders) | 33 | 58 | 64
Peripheral sensory neuropathy (Nervous system disorders) | 20 | 58 | 64
Speech disorder (Nervous system disorders) | 34 | 65 | 64
Tremor (Nervous system disorders) | 9 | 54 | 44
Agitation (Psychiatric disorders) | 3 | 27 | 17
Anxiety (Psychiatric disorders) | 15 | 50 | 41
Confusional state (Psychiatric disorders) | 32 | 57 | 59
Depression (Psychiatric disorders) | 19 | 55 | 62
Insomnia (Psychiatric disorders) | 39 | 85 | 77
Pollakiuria (Renal and urinary disorders) | 5 | 21 | 21
Urinary incontinence (Renal and urinary disorders) | 8 | 14 | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 49 | 53
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 | 35 | 37
Alopecia (Skin and subcutaneous tissue disorders) | 86 | 173 | 191
Dermatitis exfoliative NOS (Skin and subcutaneous tissue disorders) | 13 | 63 | 76
Pruritus (Skin and subcutaneous tissue disorders) | 15 | 45 | 53

LIMITATIONS AND CAVEATS:
Only participants registered after 07-12-2007 were able to participate in the quality of life / patient reported outcome study components.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No